CLINICAL TRIAL: NCT04955262
Title: A Phase 1b, Open Label, Multicenter Study of Positron Emission Tomography With Computed Tomography (PET/CT) Using ⁸⁹Zr Df-IAB22M2C (CD8 PET/CT Tracer) in Patients With Metastatic Melanoma Receiving Bempegaldesleukin (NKTR-214) and Nivolumab
Brief Title: A CD8 Positron Emission Tomography With Computed Tomography (PET/CT) Study Using ⁸⁹Zr Df-IAB22M2C in Patients With Metastatic Melanoma Receiving Bempegaldesleukin (NKTR-214) and Nivolumab
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Did not initiate due to business reasons. IND is inactive.
Sponsor: Nektar Therapeutics (Industry)
Collaborators: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-214-12
Record Dates: First submitted 2019-06-26; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Melanoma
Keywords: CD122; Immuno-oncology; Immunotherapy; Natural Killer Cells; Interleukin-2; IL-2; Nivolumab; NKTR-214; Bempegaldesleukin; Opdivo®; PD-L1; PET/CT; CD8; T-cell; Imaging; Melanoma; TIL
MeSH Terms: conditions — Melanoma | interventions — bempegaldesleukin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 Initial Cohort to Evaluate the Biodistribution of CD8 Cells (Experimental): During Cycle 1, patients will receive single-agent NKTR-214, 3 injections of 89Zr-Df-IAB22M2C, and 6 PET/CT scans. Starting with Cycle 2, patients will receive NKTR-214 in combination with nivolumab q3w for the remainder of the study. Once the PET/CT imaging data from Part 1 have been reviewed, Part 2 will open for enrollment.
  Interventions: Biological: Bempegaldesleukin (NKTR-214); Biological: Nivolumab; Drug: ⁸⁹Zr-Df-IAB22M2C
- Part 2 Expansion Cohort to Evaluate the Biodistribution of CD8 Cells (Experimental): During Cycle 1, patients will receive single-agent NKTR-214 or nivolumab, 2 injections of 89Zr-Df-IAB22M2C, and 3 PET/CT scans. In Cycle 2 and beyond, patients will receive NKTR-214 in combination with nivolumab q3w for the remainder of the study. During Cycle 2, patients will receive 1 injection of 89Zr-Df-IAB22M2C and 1 PET/CT scan.
  Interventions: Biological: Bempegaldesleukin (NKTR-214); Biological: Nivolumab; Drug: ⁸⁹Zr-Df-IAB22M2C

INTERVENTIONS:
Biological: Bempegaldesleukin (NKTR-214) — Specified dose on specified days
  Other Names: CD122-Biased Agonist; BMS-986321
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo®; BMS-936658
Drug: ⁸⁹Zr-Df-IAB22M2C — Specified dose on specified days

SUMMARY:
The main purpose of this study is to investigate the utility of the new investigational imaging agent ⁸⁹Zr Df-IAB22M2C (CD8 PET/CT tracer) to monitor CD8 T-cell expansion and trafficking within tumors and associated tissues in patients with metastatic melanoma undergoing treatment with bempegaldesleukin and nivolumab as a single agent and in combination.

DETAILED DESCRIPTION:
NKTR-214 is a cytokine (Investigational Agent), a protein which is found to expand certain immune cells (known as CD8+ T Cells and Natural Killer Cells) to promote their anti-tumor effects. Nivolumab is a full human monoclonal antibody that binds to a molecule called PD-1 (programmed cell death protein 1) on immune cells and promotes anti-tumor effects.

⁸⁹Zr Df-IAB22M2C is an experimental injected molecule containing a radioactive atom; this molecule attaches to CD8+ T cells and allows those T cells to be seen on PET/CT scans.

Part 1: A total of 4 eligible patients will be enrolled into part 1. During Cycle 1, patients will receive single agent NKTR-214, 3 injections ⁸⁹Zr Df-IAB22M2C , and 6 PET/CT scans. Starting with Cycle 2, patients will receive NKTR-214 in combination with nivolumab q3w for the remainder of the study.

Once the PET/CT imaging data from Part 1 have been reviewed, Part 2 will open for enrollment.

Part 2: A total of 20 eligible patient will be enrolled into part 2. During Cycle 1, patients will receive single agent NKTR-214 or nivolumab, 2 injections of ⁸⁹Zr Df-IAB22M2C , and 3 PET/CT scans. In Cycle 2 and beyond, patients will receive NKTR-214 in combination with nivolumab q3w for the remainder of the study. During Cycle 2, patients will receive 1 injection of ⁸⁹Zr Df-IAB22M2C and 1 PET/CT scan.

All patients enrolled in the study will be closely monitored to determine if there is response to the treatment as well as for any side effects that may occur. The efficacy of the combination will be assessed using objective response rate (ORR). Exploratory immunological biomarkers in plasma and tumor samples will evaluate immune activation.

ELIGIBILITY:
Key Inclusion Criteria:

* Provide written, informed consent to participate in the study and follow the study procedures
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1
* Measurable disease per RECIST 1.1 criteria
* Patients must have histologically confirmed metastatic melanoma with measurable, stage IV disease per American Joint Committee on Cancer (AJCC) staging system
* In patients with a single RECIST measurable lesion, the lesion must be a non-cutaneous lesion.
* Fresh biopsy
* Treatment-naive patients (i.e., no prior systemic anticancer therapy for unresectable or metastatic melanoma).

Key Exclusion Criteria:

* Patients who have an active, known or suspected autoimmune disease
* Patients must not have received prior IL-2 therapy
* Prior treatment with an anti PD-1, anti PD-L1, or anti cytotoxic T lymphocyte associated protein 4 (anti CTLA-4) antibody, agents that target IL-2, or any other antibody or drug specifically targeting T cell co-stimulation or immune checkpoint pathways
* Need for >2 antihypertensive medications for hypertension management

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Lesion uptake of 89Zr-Df-IAB22M2C (CD8 PET/CT tracer) before and after monotherapy treatment with mechanistically different immunotherapies, bempegaldesleukin (NKTR-214) and nivolumab as well as after combination treatment with NKTR-214 and nivolumab. | Approximately 18 months
  Lesion uptake of 89Zr-Df-IAB22M2C (CD8 PET/CT tracer) before and after monotherapy treatment with mechanistically different immunotherapies, bempegaldesleukin (NKTR-214) and nivolumab as well as after combination treatment with NKTR-214 and nivolumab.
Correlate ⁸⁹Zr Df-IAB22M2C lesion uptake with lesion size and ORR using PET/CT scans | Approximately 18 months
  Correlation between amount of ⁸⁹Zr Df-IAB22M2C lesion uptake (before and after monotherapy treatment and after combination treatment) with the change in lesion size and the objective response rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Nektar Therapeutics
Locations (3):
- United States (3):
  - Investigational Site - Duarte, Duarte, California
  - Investigational Site - Portland, Portland, Oregon
  - Investigational Site - Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No